CLINICAL TRIAL: NCT00655629
Title: Pivotal Phase III Trial to Investigate the Efficacy and Safety of an Orodispersible Tablet Vardenafil Versus Placebo in the Treatment of Men With Erectile Dysfunction (ED) - a Fixed-dose, Double-blind, Randomized Multi-center Trial
Brief Title: Vardenafil Orodispersible Tablet (ODT) Versus Placebo in Males With Erectile Dysfunction, 50% of Whom Are to be 65 Years or Older.
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Bayer (Industry)
Collaborators: GlaxoSmithKline (Industry); Schering-Plough (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 12094
Record Dates: First submitted 2008-04-04; First posted 2008-04-10 (Estimated); Results first posted 2011-01-21 (Estimated); Last update posted 2014-08-01 (Estimated); Status verified 2014-07

CONDITIONS: Erectile Dysfunction
Keywords: Erectile Dysfunction
MeSH Terms: conditions — Erectile Dysfunction | interventions — Vardenafil Dihydrochloride

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Vardenafil ODT (STAXYN, BAY38-9456) (Experimental): Vardenafil 10 mg orodispersible tablet (ODT) taken on demand (PRN), approximately one hour before start of sexual activity, no more than one dose per day.
  Interventions: Drug: Vardenafil ODT (STAXYN, BAY38-9456)
- Placebo (Placebo Comparator): Matching placebo tablet taken on demand (PRN), approximately one hour before start of sexual activity, no more than one dose per day.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Vardenafil ODT (STAXYN, BAY38-9456) — Subjects will receive 12 weeks of PRN (on demand) treatment with Vardenafil 10 mg orodispersible tablet (ODT)
  Arms: Vardenafil ODT (STAXYN, BAY38-9456)
Drug: Placebo — Subjects will receive 12 weeks of PRN (on demand) treatment with matching placebo tablet
  Arms: Placebo

SUMMARY:
This study investigates the safety and efficacy of a new dosage form of Vardenafil, an orodispersible tablet (ODT), and compares it to the safety and efficacy of a placebo (inactive) tablet in the treatment of erectile dysfunction. After a 4-week unmedicated phase, patients will receive Vardenafil ODT or matching placebo for 12 weeks. Safety will be determined by laboratory and other evaluations. Efficacy will be determined by the results of different questionnaires and the patient diary that will be used.

ELIGIBILITY:
Inclusion Criteria:

* Males 18 years-of-age or older.
* Stable, heterosexual relationship for at least 6 months.
* A history of erectile dysfunction (ED) for at least 6 months

Exclusion Criteria:

* Any underlying cardiovascular condition, including unstable angina pectoris
* History of myocardial infarction, stroke or life-threatening arrhythmia within 6 months prior to visit 1
* Uncontrolled atrial fibrillation / flutter at screening
* History of congenital QT prolongation
* History of surgical prostatectomy due to prostate cancer
* Hereditary degenerative retinal disorders
* History of loss of vision because of NAION (Non-arteritic anterior ischemic optic neuropathy), temporary or permanent loss of vision
* Presence of penile anatomical abnormalities
* Spinal cord injury
* Resting or postural hypotension or hypertension
* Subjects who are taking nitrates or nitric oxide donors, androgens, anti-androgens, alpha-blockers, HIV (Human immunodeficiency virus) protease inhibitors, itraconazole or ketoconazole, and clarithromycin and erythromycin.
* Subjects taking medication known to prolong QT interval, such as Type Ia and Type 3 anti-arrhythmics.
* Subjects who have been confirmed with phenylketonuria (PKU).
* Use of any treatment for ED within 7 days of Visit 1.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 339 (Actual)
Dates: Start 2008-04; Primary Completion 2009-02 (Actual); Study Completion 2009-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bayer Study Director, Study Director — Bayer
Locations (40):
- United States (21):
  - East Valley Family Physicians, PLC, Chandler, Arizona
  - Mesa Family Medical Center, Mesa, Arizona
  - Desert Clinical Research, Mesa, Arizona
  - Arizona Research Center, Inc., Phoenix, Arizona
  - Tatum Highlands Medical Associates, PLLC, Phoenix, Arizona
  - Fiel Family & Sports Medicine, PC, Tempe, Arizona
  - Irvine Center for Clinical Research, Irvine, California
  - Synergy Clinical Research Center, National City, California
  - San Diego Uro-Research, San Diego, California
  - San Diego Clinical Trials, San Diego, California
  - South Florida Medical Research, Aventura, Florida
  - Jacksonville Impotence Treatment Center, Jacksonville, Florida
  - University Clinical Research, Inc., Pembroke Pines, Florida
  - Tulane Medical Center, New Orleans, Louisiana
  - Office of Dr. Bruce Gilbert, MD, Great Neck, New York
  - Mount Sinai Medical Center, New York, New York
  - The Urology Group, Cincinnati, Ohio
  - Columbus Urology Research, LLC, Columbus, Ohio
  - Family Medical Associates, Levittown, Pennsylvania
  - Pearl Clinical Research, Norristown, Pennsylvania
  - Office of Dr. Roger Fincher, MD, Spokane, Washington
- Australia (6):
  - Sydney Men's Health, Bondi Junction, New South Wales
  - Berry Road Medical Centre, St Leonards, New South Wales
  - South Terrace Urology, Adelaide, South Australia
  - Cabrini Medical Centre, Melbourne, Victoria
  - Queen Elizabeth II Medical Centre, Nedlands, Western Australia
  - Perth Human Sexuality Centre, Perth, Western Australia
- Canada (8):
  - St.Joseph's Health Care-London, London, Ontario
  - The Male Health Centres, Oakville, Ontario
  - Office of Dr. Rajiv Singal, MD, Toronto, Ontario
  - Sunnybrook Health Sciences Centre, Toronto, Ontario
  - Clinique d'Urologie du Saguenay, Chicoutimi, Quebec
  - Urology South Shore Research, Greenfield Park, Quebec
  - Centre de Recherche en Sante Sexuelle du Quebec, Montreal, Quebec
  - Sir Mortimer B. Davis Jewish General Hospital, Montreal, Quebec
- Mexico (5):
  - Consultorio Dr. Rodríguez Rivera, Guadalajara, Jalisco
  - Hospital Dalinde, México, D. F., Mexico City
  - Centro Médico de las Américas, Mérida, Yucatán
  - Asociación Mexicana para la Salud Sexual A. C., México D. F.
  - Hospital Santa Fé, México, D. F.

REFERENCES:
- [Result] Debruyne FM, Gittelman M, Sperling H, Borner M, Beneke M. Time to onset of action of vardenafil: a retrospective analysis of the pivotal trials for the orodispersible and film-coated tablet formulations. J Sex Med. 2011 Oct;8(10):2912-23. doi: 10.1111/j.1743-6109.2011.02462.x. Epub 2011 Aug 30. PMID 21883954
- [Result] Gittelman M, McMahon CG, Rodriguez-Rivera JA, Beneke M, Ulbrich E, Ewald S. The POTENT II randomised trial: efficacy and safety of an orodispersible vardenafil formulation for the treatment of erectile dysfunction. Int J Clin Pract. 2010 Apr;64(5):594-603. doi: 10.1111/j.1742-1241.2010.02358.x. PMID 20456213

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects recruited to 35 investigational centers in the USA (20), Canada (4), Mexico (5), and Australia (6). First patient first visit on 28 Apr 2008, last patient last visit on 13 Feb 2009.
Pre-assignment Details: 473 subjects screened (<65 years: n=230; >=65 years: n=243), 339 randomized (Vardenafil 10 mg ODT=172, placebo=167). The main efficacy analysis set was the ITT (Intent to Treat) population (randomized treated sub. with baseline and post-baseline in any of the efficacy variables and safety assessment); Vardenafil 10 mg ODT=169, placebo=162
Period: Overall Study
Arm/Group | Vardenafil ODT (STAXYN, BAY38-9456) | Placebo
Started | 172 | 167
Participants Received Treatment | 171 (1 patient could not verify drug ingestion. (safety population)) | 166 (1 patient could not verify drug ingestion.(safety population))
Completed | 151 | 144
Not Completed | 21 | 23
Not completed — Adverse Event | 4 | 1
Not completed — Lack of Efficacy | 2 | 12
Not completed — Lost to Follow-up | 4 | 3
Not completed — Protocol Violation | 5 | 3
Not completed — consent withdrawn | 6 | 4

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Vardenafil ODT (STAXYN, BAY38-9456) | Placebo | Total
Number analyzed (Participants) | 171 | 166 | 337
Age, Customized [Number; unit: participants]
  <65 years | 86 | 84 | 170
  >=65 years | 85 | 82 | 167
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 171 | 166 | 337
Body Mass Index (BMI) [Mean (Standard Deviation); unit: Kilograms per square meter (kg/m^2)] | 28.9 (4.4) | 28.7 (4.2) | 28.8 (4.3)

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in International Index of Erectile Function (IIEF-EF Sub-Score) at 12 Weeks or Last Observation Carried Forward (LOCF)
Description: The primary variable was the treatment group difference from baseline to Week 12 or LOCF of the least square mean difference in the IIEF-EF domain score (Range: 1-30 ordinal. Directionality: severity of erectile dysfunction: <=10 'severe'; 11-16 'moderate'; 17-21 'mild to moderate'; 22-25 'mild'; >25 'no ED'.)
Time Frame: from baseline up to 12 weeks
Population: The primary data set was the ITT (Intent-to treat) population defined as all randomized treated subjects with baseline and post-baseline efficacy data
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Vardenafil ODT (STAXYN, BAY38-9456) | Placebo
Number analyzed (Participants) | 167 | 160
scores on a scale
  <65 years | 10.3 (7.78) | 1.7 (6.28)
  >=65 years | 6.7 (8.06) | 1.1 (6.01)
  Total | 8.5 (8.11) | 1.4 (6.14)
Statistical Analysis 1: Comparison: Vardenafil ODT (STAXYN, BAY38-9456) vs Placebo; Power adjustment for 3 primary efficacy variables (3 variables have to be significant in favor of Vardenafil to conclude efficacy). Statistical analysis applies to the total population; Test type: Superiority or Other; p < 0.0001, ANCOVA; Mean Difference (Final Values) = -6.92, 95% CI [-8.45 to -5.38]

2. Primary Outcome: Change in Percentage From Baseline in Success of Penetration (SEP2) at 12 Weeks
Description: SEP (Sexual Encounter Profile) items success rates are the percentage of all valid and successful intercourse attempts (items answered 'yes') in relation to all valid attempts. Here the SEP item refers to the ability to penetrate the partner.
Time Frame: from baseline up to 12 weeks of treatment
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: percentage of successful penetrations
Arm/Group | Vardenafil ODT (STAXYN, BAY38-9456) | Placebo
Number analyzed (Participants) | 168 | 161
percentage of successful penetrations
  <65 years | 33.2 (33.27) | 4.6 (34.12)
  >=65 years | 27.3 (37.39) | 3.0 (33.33)
  Total | 30.2 (35.40) | 3.8 (33.63)
Statistical Analysis 1: Comparison: Vardenafil ODT (STAXYN, BAY38-9456) vs Placebo; Statistical analysis applies to the total population; Test type: Superiority or Other; p < 0.0001, ANCOVA; Mean Difference (Final Values) = -25.972, 95% CI [-32.688 to -19.256]

3. Primary Outcome: Change From Baseline in Success of Erection Maintenance at 12 Weeks
Description: SEP items success rates are the percentage of all valid and successful intercourse attempts (items answered 'yes') in relation to all valid attempts. Here the SEP item refers to the ability to maintain an erection after penetration.
Time Frame: from baseline up to 12 weeks of treatment
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: percentage of successful maintenance
Arm/Group | Vardenafil ODT (STAXYN, BAY38-9456) | Placebo
Number analyzed (Participants) | 168 | 160
percentage of successful maintenance
  <65 years | 53.2 (33.22) | 15.2 (29.55)
  >=65 years | 38.8 (38.32) | 8.7 (29.15)
  Total | 46.0 (36.47) | 12.0 (29.44)
Statistical Analysis 1: Comparison: Vardenafil ODT (STAXYN, BAY38-9456) vs Placebo; Statistical analysis applies to the total population; Test type: Superiority or Other; p < 0.0001, ANCOVA; Mean Difference (Final Values) = -33.432, 95% CI [-40.439 to -26.425]

4. Secondary Outcome: Percentage of Subjects Achieving "Back to Normal" Erectile Function
Description: Responders: percentage of subjects achieving an IIEF-EF score > 25. The primary variable was the treatment group difference from baseline to Week 12 or Last observation carried forward (LOCF) of the least square mean difference in the IIEF-EF domain score (1-30 ordinal points, specifying the severity of erectile dysfunction: <=10 'severe'; 11-16 'moderate'; 17-21 'mild to moderate'; 22-25 'mild'; >25 'no ED').
Time Frame: up to 12 weeks of treatment
Population: as for outcome 1
Measure: Number; unit: percentage of subjects
Arm/Group | Vardenafil ODT (STAXYN, BAY38-9456) | Placebo
Number analyzed (Participants) | 167 | 160
percentage of subjects
  <65 years | 59 | 11
  >=65 years | 32 | 8
  Total | 46 | 9
Statistical Analysis 1: Comparison: Vardenafil ODT (STAXYN, BAY38-9456) vs Placebo; Statistical analysis applies to the total population; Test type: Superiority or Other; p < 0.0001, Cochran-Mantel-Haenszel; CMH adjusted for age group and center; Cochran-Mantel-Haenszel = 53.8693

5. Secondary Outcome: Change in Percentage From Baseline in Ability to Obtain an Erection at 12 Weeks
Description: SEP items success rates are the percentage of all valid and successful intercourse attempts (items answered 'yes') in relation to all valid attempts. Here the SEP item refers to the ability to obtain successful erections.
Time Frame: from baseline up to 12 weeks of treatment
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: percentage of successful erections
Arm/Group | Vardenafil ODT (STAXYN, BAY38-9456) | Placebo
Number analyzed (Participants) | 168 | 161
percentage of successful erections
  <65 years | 13.4 (28.63) | -5.8 (38.18)
  >=65 years | 9.6 (35.96) | -3.8 (37.04)
  Total | 11.5 (32.46) | -4.8 (37.51)
Statistical Analysis 1: Comparison: Vardenafil ODT (STAXYN, BAY38-9456) vs Placebo; Statistical analysis applies to the total population; Test type: Superiority or Other; p < 0.0001, ANCOVA; Mean Difference (Final Values) = -16.078, 95% CI [-22.41 to -9.746]

6. Secondary Outcome: Change in Percentage From Baseline in Satisfaction With the Hardness of Erection at 12 Weeks
Description: SEP items success rates are the percentage of all valid and successful intercourse attempts (items answered 'yes') in relation to all valid attempts. Here the SEP item refers to the ability to get satisfactory hardness of erections.
Time Frame: from baseline up to 12 weeks of treatment
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: percentage of satisfactory erections
Arm/Group | Vardenafil ODT (STAXYN, BAY38-9456) | Placebo
Number analyzed (Participants) | 168 | 160
percentage of satisfactory erections
  <65 years | 52.0 (40.04) | 12.2 (30.89)
  >=65 years | 36.1 (41.54) | 5.4 (31.21)
  Total | 44.1 (41.45) | 8.8 (31.14)
Statistical Analysis 1: Comparison: Vardenafil ODT (STAXYN, BAY38-9456) vs Placebo; Statistical analysis applies to the total population; Test type: Superiority or Other; p < 0.0001, ANCOVA; Mean Difference (Final Values) = -33.134, 95% CI [-40.281 to -25.987]

7. Secondary Outcome: Change in Percentage From Baseline in Overall Satisfaction at 12 Weeks
Description: SEP items success rates are the percentage of all valid and successful intercourse attempts (items answered 'yes') in relation to all valid attempts. Here the SEP item refers to overall satisfactory attempts.
Time Frame: from baseline up to 12 weeks of treatment
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: percentage of satisfactory attempts
Arm/Group | Vardenafil ODT (STAXYN, BAY38-9456) | Placebo
Number analyzed (Participants) | 168 | 160
percentage of satisfactory attempts
  <65 years | 52.0 (40.04) | 12.2 (30.89)
  >=65 years | 38.4 (38.43) | 10.3 (26.70)
  Total | 45.1 (40.15) | 11.2 (26.39)
Statistical Analysis 1: Comparison: Vardenafil ODT (STAXYN, BAY38-9456) vs Placebo; Statistical analysis applies to the total population; Test type: Superiority or Other; p < 0.0001, ANCOVA; Mean Difference (Final Values) = -33.934, 95% CI [-41.119 to -26.749]

8. Secondary Outcome: Change in Percentage From Baseline in Ability to Ejaculate at 12 Weeks
Description: SEP items success rates are the percentage of all valid and successful intercourse attempts (items answered 'yes') in relation to all valid attempts. Here the SEP item refers to the ability to have successful ejaculations.
Time Frame: from baseline up to 12 weeks of treatment
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: percentage of ejaculation successes
Arm/Group | Vardenafil ODT (STAXYN, BAY38-9456) | Placebo
Number analyzed (Participants) | 168 | 160
percentage of ejaculation successes
  <65 years | 37.3 (32.52) | 7.1 (35.0)
  >=65 years | 17.7 (36.27) | 2.7 (36.51)
  Total | 27.5 (35.72) | 4.9 (35.71)
Statistical Analysis 1: Comparison: Vardenafil ODT (STAXYN, BAY38-9456) vs Placebo; Statistical analysis applies to the total population; Test type: Superiority or Other; p < 0.0001, ANCOVA; Mean Difference (Final Values) = -20.902, 95% CI [-27.724 to -14.081]

9. Secondary Outcome: Number of Sexual Attempts Till First Successful Attempt
Time Frame: up to 12 weeks of treatment
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Sexual Attempts
Arm/Group | Vardenafil ODT (STAXYN, BAY38-9456) | Placebo
Number analyzed (Participants) | 134 | 92
Sexual Attempts
  <65 years | 1.2 (3.7) | 2.6 (3.5)
  >=65 years | 1.6 (4.5) | 3.8 (3.9)
  Total | 1.4 (4.1) | 3.1 (3.7)

10. Secondary Outcome: Change From Baseline in Ease With Erection at 12 Weeks or LOCF
Description: Treatment group difference in points on the Treatment Satisfaction Scale (TSS: 0-100 normalized, ordinal; Directionality: Higher scores indicate greater levels of (i) ease with erection, (ii) erectile functioning satisfaction, (iii) pleasure of sexual activity, (iv) satisfaction with orgasm, (v) confidence for completion, and (vi) satisfaction with medication.) domain "Ease with Erection" from baseline to Week 12 or LOCF expressed as the least square mean difference.
Time Frame: from baseline up to 12 weeks
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Vardenafil ODT (STAXYN, BAY38-9456) | Placebo
Number analyzed (Participants) | 158 | 158
scores on a scale
  <65 years | 24.0 (34.29) | 6.1 (31.77)
  >=65 years | 14.4 (29.17) | 0.0 (27.84)
  Total | 19.1 (32.07) | 3.0 (29.91)
Statistical Analysis 1: Comparison: Vardenafil ODT (STAXYN, BAY38-9456) vs Placebo; Statistical analysis applies to the total population; Test type: Superiority or Other; p < 0.0001, ANCOVA; Mean Difference (Final Values) = -16.866, 95% CI [-22.599 to -11.133]

11. Secondary Outcome: Change From Baseline in Erectile Function Satisfaction at 12 Weeks or LOCF
Description: Treatment group difference in points on the Treatment Satisfaction Scale (TSS: 0-100 normalized, ordinal; Directionality: Higher scores indicate greater levels of (i) ease with erection, (ii) erectile functioning satisfaction, (iii) pleasure of sexual activity, (iv) satisfaction with orgasm, (v) confidence for completion, and (vi) satisfaction with medication.) domain "Erectile function satisfaction" from baseline to Week 12 or LOCF expressed as the least square mean difference
Time Frame: from baseline up to 12 weeks
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Vardenafil ODT (STAXYN, BAY38-9456) | Placebo
Number analyzed (Participants) | 158 | 158
scores on a scale
  <65 years | 41.2 (27.78) | 7.6 (24.95)
  >=65 years | 25.4 (26.11) | 4.2 (24.84)
  Total | 33.2 (28.01) | 5.9 (24.88)
Statistical Analysis 1: Comparison: Vardenafil ODT (STAXYN, BAY38-9456) vs Placebo; Statistical analysis applies to the total population; Test type: Superiority or Other; p < 0.0001, ANCOVA; Mean Difference (Final Values) = -26.040, 95% CI [-31.547 to -20.533]

12. Secondary Outcome: Change From Baseline in Pleasure of Sexual Activity at 12 Weeks or LOCF
Description: Treatment group difference in points on the Treatment Satisfaction Scale (TSS: 0-100 normalized, ordinal; Directionality: Higher scores indicate greater levels of (i) ease with erection, (ii) erectile functioning satisfaction, (iii) pleasure of sexual activity, (iv) satisfaction with orgasm, (v) confidence for completion, and (vi) satisfaction with medication.) domain "Pleasure of sexual activity" from baseline to Week 12 or LOCF expressed as the least square mean difference
Time Frame: from baseline up to 12 weeks
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Vardenafil ODT (STAXYN, BAY38-9456) | Placebo
Number analyzed (Participants) | 158 | 158
scores on a scale
  <65 years | 30.1 (24.63) | 4.8 (25.82)
  >=65 years | 15.3 (29.63) | -1.9 (22.42)
  Total | 22.6 (28.19) | 1.4 (24.31)
Statistical Analysis 1: Comparison: Vardenafil ODT (STAXYN, BAY38-9456) vs Placebo; Statistical analysis applies to the total population; Test type: Superiority or Other; p < 0.0001, ANCOVA; Mean Difference (Final Values) = -19.496, 95% CI [-24.676 to -14.315]

13. Secondary Outcome: Change From Baseline in Satisfaction With Orgasm at 12 Weeks or LOCF
Description: Treatment group difference in points on the Treatment Satisfaction Scale (TSS: 0-100 normalized, ordinal; Directionality: Higher scores indicate greater levels of (i) ease with erection, (ii) erectile functioning satisfaction, (iii) pleasure of sexual activity, (iv) satisfaction with orgasm, (v) confidence for completion, and (vi) satisfaction with medication.) domain "Satisfaction with orgasm" from baseline to Week 12 or LOCF expressed as the least square mean difference
Time Frame: from baseline up to 12 weeks
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Vardenafil ODT (STAXYN, BAY38-9456) | Placebo
Number analyzed (Participants) | 158 | 157
scores on a scale | 23.6 (30.81) | 3.2 (31.36)
Statistical Analysis 1: Comparison: Vardenafil ODT (STAXYN, BAY38-9456) vs Placebo; Statistical analysis applies to the total population; Test type: Superiority or Other; p < 0.0001, ANCOVA; Mean Difference (Final Values) = -18.418, 95% CI [-24.439 to -12.396]

14. Secondary Outcome: Change From Baseline in Confidence for Completion at 12 Weeks or LOCF
Description: Treatment group difference in points on the Treatment Satisfaction Scale (TSS: 0-100 normalized, ordinal; Directionality: Higher scores indicate greater levels of (i) ease with erection, (ii) erectile functioning satisfaction, (iii) pleasure of sexual activity, (iv) satisfaction with orgasm, (v) confidence for completion, and (vi) satisfaction with medication.) domain "Confidence for completion" from baseline to Week 12 or LOCF expressed as the least square mean difference
Time Frame: from baseline up to 12 weeks
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Vardenafil ODT (STAXYN, BAY38-9456) | Placebo
Number analyzed (Participants) | 158 | 158
scores on a scale
  <65 years | 38.0 (28.59) | 4.8 (28.22)
  >=65 years | 20.2 (27.74) | 2.8 (27.05)
  Total | 29.0 (29.46) | 3.8 (27.56)
Statistical Analysis 1: Comparison: Vardenafil ODT (STAXYN, BAY38-9456) vs Placebo; Statistical analysis applies to the total population; Test type: Superiority or Other; p < 0.0001, ANCOVA; Mean Difference (Final Values) = -22.379, 95% CI [-28.006 to -16.753]

15. Secondary Outcome: Satisfaction With Medication at Week 12 or LOCF
Description: Treatment group difference in points on the Treatment Satisfaction Scale (TSS: 0-100 normalized, ordinal; Directionality: Higher scores indicate greater levels of (i) ease with erection, (ii) erectile functioning satisfaction, (iii) pleasure of sexual activity, (iv) satisfaction with orgasm, (v) confidence for completion, and (vi) satisfaction with medication.) domain "Satisfaction with medication" at LOCF expressed as the least square mean difference
Time Frame: up to 12 weeks
Population: The primary data set was the ITT (Intent-to treat) population defined as all randomized treated subjects with LOCF values.
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Vardenafil ODT (STAXYN, BAY38-9456) | Placebo
Number analyzed (Participants) | 159 | 158
scores on a scale
  <65 years | 58.6 (26.55) | 19.3 (26.55)
  >=65 years | 42.5 (30.26) | 20.2 (24.59)
  Total | 50.5 (29.52) | 19.7 (25.50)
Statistical Analysis 1: Comparison: Vardenafil ODT (STAXYN, BAY38-9456) vs Placebo; Statistical analysis applies to the total population; Test type: Superiority or Other; p < 0.0001, ANOVA; Mean Difference (Final Values) = -30.758, 95% CI [-36.736 to -24.779]

16. Secondary Outcome: Patient Self Reported Improvement of Erectile Function Under Treatment Using a Categorical Rating Scale
Description: Categorical Rating Scale is a binary rating scale with 2 response options which is 'yes/no'; percentage of participants with positive answers to the Global Assessment Question. Global Assessment Question (GAQ): 'Has the treatment you have been taking over the past for weeks improved your erection?' (yes/no)
Time Frame: up to 12 weeks of treatment
Population: as for outcome 1
Measure: Number; unit: percentage of participants
Arm/Group | Vardenafil ODT (STAXYN, BAY38-9456) | Placebo
Number analyzed (Participants) | 160 | 157
percentage of participants
  <65 years | 75 | 19
  >=65 years | 59 | 28
  Total | 67 | 24
Statistical Analysis 1: Comparison: Vardenafil ODT (STAXYN, BAY38-9456) vs Placebo; Statistical analysis applies to the total population; Test type: Superiority or Other; p < 0.0001, Cochran-Mantel-Haenszel; CMH adjusted for age group and center; Cochran-Mantel-Haenszel = 60.2391

ADVERSE EVENTS:
Arm/Group | Vardenafil ODT (STAXYN, BAY38-9456) | Placebo
Serious Adverse Events (participants affected / at risk) | 2/171 | 1/166
Other Adverse Events (participants affected / at risk) | 65/171 | 37/166
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Vardenafil ODT (STAXYN, BAY38-9456) (N=171) | Placebo (N=166)
Arrhythmia (Cardiac disorders) | 1 | 0
Chest pain (General disorders) | 1 | 0
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Hypertension (Vascular disorders) | 1 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Vardenafil ODT (STAXYN, BAY38-9456) (N=171) | Placebo (N=166)
Bundle branch block (Cardiac disorders) | 1 | 0
Bundle branch block right (Cardiac disorders) | 0 | 1
Mitral valve incompetence (Cardiac disorders) | 1 | 0
Supraventricular extrasystoles (Cardiac disorders) | 1 | 1
Tricuspid valve incompetence (Cardiac disorders) | 1 | 0
Ventricular extrasystoles (Cardiac disorders) | 2 | 2
Left ventricular hypertrophy (Cardiac disorders) | 1 | 0
Vertigo (Ear and labyrinth disorders) | 1 | 0
Diplopia (Eye disorders) | 1 | 0
Eye pain (Eye disorders) | 1 | 0
Vision blurred (Eye disorders) | 1 | 1
Eye pruritus (Eye disorders) | 1 | 0
Abdominal pain (Gastrointestinal disorders) | 0 | 1
Abdominal pain upper (Gastrointestinal disorders) | 1 | 0
Colonic polyp (Gastrointestinal disorders) | 0 | 1
Constipation (Gastrointestinal disorders) | 0 | 1
Diarrhoea (Gastrointestinal disorders) | 3 | 1
Dry mouth (Gastrointestinal disorders) | 2 | 1
Dyspepsia (Gastrointestinal disorders) | 3 | 0
Dysphagia (Gastrointestinal disorders) | 1 | 0
Nausea (Gastrointestinal disorders) | 1 | 0
Toothache (Gastrointestinal disorders) | 1 | 0
Chest discomfort (General disorders) | 1 | 0
Chest pain (General disorders) | 2 | 0
Fatigue (General disorders) | 1 | 0
Feeling hot (General disorders) | 1 | 0
Pyrexia (General disorders) | 1 | 0
Influenza (Infections and infestations) | 1 | 0
Nasopharyngitis (Infections and infestations) | 0 | 3
Pharyngitis (Infections and infestations) | 3 | 3
Pharyngitis streptococcal (Infections and infestations) | 0 | 1
Pneumonia (Infections and infestations) | 1 | 0
Rhinitis (Infections and infestations) | 2 | 0
Sinusitis (Infections and infestations) | 1 | 2
Tooth abscess (Infections and infestations) | 0 | 2
Upper respiratory tract infection (Infections and infestations) | 3 | 0
Urinary tract infection (Infections and infestations) | 1 | 0
Bacterial rhinitis (Infections and infestations) | 1 | 0
Arthropod sting (Injury, poisoning and procedural complications) | 0 | 1
Multiple injuries (Injury, poisoning and procedural complications) | 1 | 0
Muscle injury (Injury, poisoning and procedural complications) | 1 | 0
Contusion (Injury, poisoning and procedural complications) | 1 | 0
Penis deviation (Injury, poisoning and procedural complications) | 1 | 0
Arthroscopy (Investigations) | 0 | 1
Blood creatinine increased (Investigations) | 1 | 0
Blood pressure increased (Investigations) | 2 | 0
Cardiac murmur (Investigations) | 1 | 0
Heart rate increased (Investigations) | 1 | 0
Diabetes mellitus (Metabolism and nutrition disorders) | 1 | 1
Gout (Metabolism and nutrition disorders) | 1 | 0
Hypertriglyceridaemia (Metabolism and nutrition disorders) | 1 | 0
Hyperlipidaemia (Metabolism and nutrition disorders) | 1 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 4 | 1
Joint swelling (Musculoskeletal and connective tissue disorders) | 1 | 0
Muscle spasms (Musculoskeletal and connective tissue disorders) | 2 | 0
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1 | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 1 | 0
Neck pain (Musculoskeletal and connective tissue disorders) | 2 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 | 0
Spinal osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 | 0
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Burning sensation (Nervous system disorders) | 1 | 0
Dizziness (Nervous system disorders) | 5 | 0
Headache (Nervous system disorders) | 21 | 4
Sinus headache (Nervous system disorders) | 1 | 0
Anxiety (Psychiatric disorders) | 0 | 1
Prostatitis (Reproductive system and breast disorders) | 0 | 1
Testicular pain (Reproductive system and breast disorders) | 0 | 1
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 8 | 1
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Sleep apnoea syndrome (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Wheezing (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 1 | 0
Ingrowing nail (Skin and subcutaneous tissue disorders) | 0 | 1
Night sweats (Skin and subcutaneous tissue disorders) | 1 | 0
Rash (Skin and subcutaneous tissue disorders) | 2 | 2
Pharmaceutical product complaint (Social circumstances) | 0 | 1
Skin lesion excision (Surgical and medical procedures) | 0 | 1
Cataract operation (Surgical and medical procedures) | 1 | 0
Flushing (Vascular disorders) | 13 | 2
Hypertension (Vascular disorders) | 1 | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
In the protocol it is specified that all results are the property of the sponsor. The investigator must discuss any publication with the sponsor prior to release and obtain written consent of the sponsor. The investigator must send a draft publication to the sponsor thirty days in advance of submission in order to obtain approval prior to submission of the final version for publication.